CLINICAL TRIAL: NCT00445133
Title: A Double-Blind, Randomized, Placebo-Controlled Study on Magnetic Field Therapy to Improve Quality of Sleep and Reduction of Chronic Spine Pain (Sleep/Mag)
Brief Title: Study on Magnetic Field Therapy to Improve Quality of Sleep and Reduction of Chronic Spine Pain
Acronym: SLEEP/MAG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00781440
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Back Pain; Neck Pain; Sleep Initiation and Maintenance Disorders
Keywords: Neck Pain/Lumbar pain/Magnets/sleep deficiency/ insomnia/
MeSH Terms: conditions — Back Pain; Neck Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magnetic Sleep Pad

SUMMARY:
HYPTHOTHESIS:

The researchers hypothesize that application of active magnetic therapy vs. sham utilized while individuals sleep can reduce neuropathic pain in the spine and improve the quality of sleep. The null hypothesis is that treatment of subjects with spine pain with exposure to permanent/static magnetic fields has no measurable effect on neuropathic pain scores or quality of sleep scores.

DETAILED DESCRIPTION:
DESIGN:

This is a double-blind, randomized, placebo-controlled study which will consist of two treatment groups. Treated subjects will receive a permanent/static magnetic sleeping pad with a nominal strength of less than 1000 Gauss. Control subjects will receive physically identical sleeping pad with a nominal surface field strength of 0 Gauss (placebo). The magnets will be contained in a standard mattress pad and subjects will sleep on the pad. The primary outcome measures will be quality of sleep as well as the daily VAS scores. These are subjective. There will be objective assessment by the quantification of autonomic nervous system (ANS) strengths of the parasympathetic and sympathetic effects from this non-invasive digital study using spectral analysis. Individuals will be evaluated at onset of study and at end of study to look at specifics of range of motion, spasm, radiculitis, etc. Scores will be kept on a monthly basis as well as repeat of ANS testing each month. At the end of the study, individuals will return all forms, be reevaluated by Dr. Weintraub and also will be asked questions regarding PGIC for bias, etc. Additionally heart rate and systolic and diastolic BP readings at rest and with challenge of standing will be recorded at baseline and each visit to determine if there is an anti-hypertensive effect from sleeping on magnetic device. A reduction of 3 mm Hg improves stroke and cardiac risk by a minimum of 4%. No new anti-hypertensive medications will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects age 18-80.
* Capable of understanding and complying with study protocols.
* Chronic cervical, thoracic or lumbar pain for at least six months.
* Sleep difficulties and/or insomnia

Exclusion Criteria:

* Unable to understand informed consent (mental retardation, psychosis, communicative impairment).
* Cardiac pacemaker or other mechanical internal devices.
* Tumor in the spine/history of malignancy.
* Pregnancy.
* Prior spine surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-02; Study Completion 2007-12

PRIMARY OUTCOMES:
VAS Pain scores/Pittsburgh Sleep scores/Insomnia sleep scores/SF 15 pain descriptor scores/PGIC/

SECONDARY OUTCOMES:
Autonomic Nerve Functions

CONTACTS AND LOCATIONS:
Overall Officials: Michael I. Weintraub, MD, Principal Investigator — Phelps Memorial Hospital
Locations (1):
- Dr. Michael I . Weintraub, Briarcliff Manor, New York, United States